CLINICAL TRIAL: NCT01717326
Title: A Phase II Randomized Clinical Trial to Study the Efficacy and Safety of the Combination Regimen MK-5172 and MK-8742 ± Ribavirin (RBV) in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: A Study of the Combination Regimen Grazoprevir (MK-5172) and Elbasvir (MK-8742) ± Ribavirin in Participants With Chronic Hepatitis C (MK-5172-035)
Acronym: C-WORTHy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-035; 2012-003354-89 (EudraCT Number)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (20):
- A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk (Experimental): GT1a and GT1b participants receive Grazoprevir 100 mg tablet orally once daily (QD) for 12 weeks, Elbasvir 20 mg capsule and Placebo capsule orally QD for 12 weeks, RBV capsules orally twice daily (BID) for 24 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Placebo to Elbasvir; Drug: Ribavirin
- A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (Experimental): GT1a and GT1b participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule and Placebo capsule orally QD for 12 weeks, RBV capsules orally BID for 24 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Placebo to Elbasvir; Drug: Ribavirin
- A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg-12 wk (Experimental): GT1b only participants receive Grazoprevr 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (Experimental): GT1a only participants receive Grazoprevir 100 mg tablet orally QD for 8 weeks, Elbasvir 50 mg capsule orally QD for 8 weeks, RBV capsules orally BID for 8 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg-12 wk (Experimental): GT1a only participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 18 weeks, Elbasvir 50 mg capsule orally QD for 18 weeks, RBV capsules orally BID for 18 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B7: TN C Grazoprevir 100 mg + Elbasvir 50 mg-18 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 18 weeks, Elbasvir 50 mg capsule orally QD for 18 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B9: NR Grazoprevir 100 mg + Elbasvir 50 mg-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 18 weeks, Elbasvir 50 mg capsule orally QD for 18 weeks, RBV capsules orally BID for 18 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B11: NR Grazoprevir 100 mg + Elbasvir 50 mg-18 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 18 weeks, Elbasvir 50 mg capsule orally QD for 18 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg-12 wk (Experimental): GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (Experimental): GT1b participants receive Grazoprevir 100 mg tablet orally QD for 8 weeks, Elbasvir 50 mg capsule orally QD for 8 weeks, and RBV capsules orally BID for 8 weeks at a total daily dose from 800 to 1400 mg based on participant weight.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg-8 wk (Experimental): GT1b participants receive Grazoprevir 100 mg tablet orally QD for 8 weeks and Elbasvir 50 mg capsule orally QD for 8 weeks
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (Experimental): GT3 participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, and RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin
- D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (Experimental): GT3 participants receive Grazoprevir 100 mg tablet orally QD for 18 weeks, Elbasvir 50 mg capsule orally QD for 18 weeks, and RBV capsules orally BID for 18 weeks at a total daily dose from 800 to 1400 mg based on participant weight
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Grazoprevir — 100 mg tablet orally QD
  Other Names: MK-5172
Drug: Elbasvir — Part A: 20 or 50 mg capsule orally QD Parts B, C, and D: 50 mg capsule orally QD
  Other Names: MK-8742
Drug: Placebo to Elbasvir — Placebo to Elbasvir 20 or 50 mg capsule, orally, once daily for 12 weeks to maintain blind (Part A only)
  Arms: A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk; A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk
Drug: Ribavirin — Oral capsules BID at a total daily dose from 800 to 1400 mg based on participant weight
  Other Names: Rebetol™; RBV
  Arms: A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk; A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk; B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk; B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk; B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk; C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk; D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk

SUMMARY:
This is a study of the safety and efficacy of grazoprevir (MK-5172) in combination with elbasvir (MK-8742) ± ribavirin (RBV). The primary efficacy endpoint will be Sustained Virologic Response 12 weeks after the end of all study therapy (SVR12) in each of the treatment arms.

DETAILED DESCRIPTION:
Part A is being done in treatment-naïve (TN), genotype 1 (GT1), interferon eligible, non-cirrhotic (N-C) participants with chronic hepatitis C (CHC). Participants will be assigned randomly to 1 of 2 treatment arms in which they will receive grazoprevir 100 mg once daily (QD) + elbasvir 20 mg or 50 mg QD and twice daily (BID) RBV, or to a treatment arm in which they will receive grazoprevir 100 mg QD + elbasvir 50 mg QD without RBV. Treatment will last 12 weeks.

In Part B, participants with hepatitis C virus (HCV) GT1 and HCV ribonucleic acid (RNA) levels of ≥10,000 IU/mL will be randomly assigned to a study arm, based on absence or presence of cirrhosis (C), whether they are TN or had poor response to previous antiviral therapy (null responders [NR]), or whether co-infected with human immunodeficiency virus (HIV); these participants will receive open-label grazoprevir (100 mg) in combination with elbasvir (50 mg) ± RBV. Treatment will last 8 to 18 weeks dependent on arm assignment.

In Part C, TN, N-C participants with HCV GT1b and HCV RNA levels of ≥10,000 IU/mL will be randomly assigned to receive open-label grazoprevir (100 mg) in combination with elbasvir (50 mg) ± RBV. Treatment will last 8 weeks.

In Part D, TN N-C participants with HCV GT3 and HCV RNA levels of ≥10,000 IU/mL will be randomly assigned to receive open-label grazoprevir (100 mg) in combination with elbasvir (50 mg) + RBV for 12 or 18 weeks.

ELIGIBILITY:
Inclusion criteria:

All participants

* CHC genotype 1 (GT1) virus infection (Parts A, B, and C) or GT3 virus infection (Part D)
* Female participants of childbearing potential or male participant with female partners of childbearing potential, must use two acceptable methods of birth control from ≥2 weeks prior to Day 1 until ≥6 months after last dose of study drug, or longer if dictated by local regulations

Part A - Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease, or cirrhosis - No evidence of advanced fibrosis, cirrhosis and/or hepatocellular carcinoma by biopsy or noninvasive testing (FibroScan and/or FibroTest)

Parts B, C, and D

* Treatment naïve with or without cirrhosis, or
* Prior treatment failure to Peg-IFN/Ribavirin with or without cirrhosis, or
* Co-infected with human immunodeficiency virus (HIV) without cirrhosis
* Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease
* Liver disease staging assessment by liver biopsy or noninvasive testing (FibroScan and/or FibroTest)

Exclusion criteria:

All participants

* Non-GT1 HCV infection (Part A, Part B, and Part C) or a non-GT3 HCV infection (Part D) including a mixed GT infection (with a non-GT1 [Part A, Part B, and Part C] or non-GT3 [Part D]) or a non-typeable genotype
* Evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Currently participating or participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another study
* Diabetic and/or hypertensive with clinically significant ocular examination findings
* History of depression associated with hospitalization for depression, electroconvulsive therapy, or resulting in prolonged absence from work and/or significant disruption of daily functions
* Suicidal or homicidal ideations and/or attempt, or history of severe psychiatric disorders
* Clinical diagnosis of substance abuse
* Current history of seizure disorder, stroke, or transient ischemic attack
* Immunologically mediated disease
* Chronic pulmonary disease
* Clinically significant cardiac abnormalities/dysfunction
* Active clinical gout within the last year
* Hemoglobinopathy or myelodysplastic syndromes
* History of organ transplants including hematopoietic stem cell transplants
* Poor venous access
* Indwelling venous catheter
* History of gastric surgery or malabsorption disorders
* Severe concurrent disease
* Evidence of active or suspected malignancy, or a history of malignancy, ≤5 years before
* Pregnant, lactating, expecting to conceive or donate eggs
* Male participant with pregnant female partner
* Member/family member of the investigational study or sponsor staff directly involved with this study
* Evidence or history of chronic hepatitis not caused by HCV

Part A

* Not treatment-naïve
* Documented to be HIV positive
* Taking or planning to take significant inducers or inhibitors of CYP3A4 substrates or herbal supplements 2 weeks prior to start of study medications

Parts B, C, and D

* Previously received any HCV direct-acting antivirals
* Requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* For participants diagnosed with diabetes mellitus, documented HbA1c >8.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2013-02-07 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-05-06 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Lawitz E, Gane E, Pearlman B, Tam E, Ghesquiere W, Guyader D, Alric L, Bronowicki JP, Lester L, Sievert W, Ghalib R, Balart L, Sund F, Lagging M, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 12 weeks versus 18 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin for hepatitis C virus genotype 1 infection in previously untreated patients with cirrhosis and patients with previous null response with or without cirrhosis (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1075-86. doi: 10.1016/S0140-6736(14)61795-5. Epub 2014 Nov 11. PMID 25467591
- [Background] Sulkowski M, Hezode C, Gerstoft J, Vierling JM, Mallolas J, Pol S, Kugelmas M, Murillo A, Weis N, Nahass R, Shibolet O, Serfaty L, Bourliere M, DeJesus E, Zuckerman E, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 8 weeks versus 12 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin in patients with hepatitis C virus genotype 1 mono-infection and HIV/hepatitis C virus co-infection (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1087-97. doi: 10.1016/S0140-6736(14)61793-1. Epub 2014 Nov 11. PMID 25467560
- [Derived] Gane E, Nahass R, Luketic V, Asante-Appiah E, Hwang P, Robertson M, Wahl J, Barr E, Haber B. Efficacy of 12 or 18 weeks of elbasvir plus grazoprevir with ribavirin in treatment-naive, noncirrhotic HCV genotype 3-infected patients. J Viral Hepat. 2017 Oct;24(10):895-899. doi: 10.1111/jvh.12719. Epub 2017 Jun 23. PMID 28470815
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male/female participants with Hepatitis C Virus (HCV) genotype 1 (GT1) or GT3 who were either treatment-naïve (TN) or prior null responder (NR), cirrhotic (C) or noncirrhotic (NC), and monoinfected with HCV or coinfected with HCV and human immunodeficiency virus (HIV) were recruited based on entry requirements for Parts A, B, C, or D.
Pre-assignment Details: 573 participants were randomized on study. 65 TN NC GT1 participants were randomized in Part A. Part B randomized 94 TN NC participants, 123 TN C participants, 130 NR participants (C and NC), and 59 TN HIV coinfected participants. Part C randomized 61 TN NC GT1b participants, and Part D randomized 41 TN NC GT3 participants.
Groups:
- B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk; B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk; B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk: GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 12 weeks, Elbasvir 50 mg capsule orally QD for 12 weeks, RBV capsules orally BID for 12 weeks at a total daily dose from 800 to 1400 mg based on participant weight.
- B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk: GT1a/non-a participants receive Grazoprevir 100 mg tablet orally QD for 8 weeks, Elbasvir 50 mg capsule orally QD for 8 weeks, RBV capsules orally BID for 8 weeks at a total daily dose from 800 to 1400 mg based on participant weight.
Period: Overall Study
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Started | 25 | 27 | 13 | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21
Treated | 25 | 28 (Number includes 1 additional participant randomized to A3 but treated on A2) | 12 (Number excludes 1 participant randomized to A3 but treated on Arm A2) | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21
Completed | 22 | 26 | 13 | 28 | 31 | 31 | 30 | 29 | 32 | 29 | 30 | 33 | 32 | 32 | 29 | 27 | 29 | 31 | 16 | 15
Not Completed | 3 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 4 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS); all randomized participants who received ≥1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | Total
Number analyzed (Participants) | 25 | 27 | 13 | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.5) | 43.9 (12.6) | 43.3 (13.5) | 48.4 (11.9) | 49.7 (11.5) | 53.6 (8.4) | 57.0 (7.0) | 59.0 (7.8) | 58.8 (8.2) | 58.9 (8.0) | 52.2 (8.8) | 54.4 (9.1) | 56.2 (10.9) | 54.3 (12.3) | 46.2 (8.4) | 43.5 (10.4) | 50.6 (10.9) | 55.3 (10.3) | 49.0 (11.5) | 42.4 (10.8) | 51.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 6 | 12 | 15 | 15 | 12 | 10 | 17 | 10 | 12 | 13 | 17 | 14 | 6 | 6 | 14 | 18 | 12 | 13 | 252
  Male | 12 | 10 | 7 | 18 | 18 | 16 | 19 | 19 | 15 | 21 | 20 | 20 | 16 | 18 | 23 | 24 | 16 | 13 | 8 | 8 | 321

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of All Study Therapy (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). SVR12 was defined as HCV RNA <25 IU/ml at 12 weeks after the end of all study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: 12 weeks after end of therapy (up to 30 weeks)
Population: The Per-Protocol (PP) population; all randomized participants who received ≥1 dose of study treatment and without important protocol deviations who had data available at the respective time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 22 | 24 | 12 | 29 | 29 | 31 | 30 | 29 | 31 | 31 | 30 | 33 | 33 | 32 | 29 | 28 | 29 | 31 | 19 | 18
percentage of participants | 100.0 [84.6 to 100.0] | 95.8 [78.9 to 99.9] | 100.0 [73.5 to 100.0] | 82.8 [64.2 to 94.2] | 100.0 [88.1 to 100.0] | 96.8 [83.3 to 99.9] | 90.0 [73.5 to 97.9] | 96.6 [82.2 to 99.9] | 100.0 [88.8 to 100.0] | 93.5 [78.6 to 99.2] | 100.0 [88.4 to 100.0] | 90.9 [75.7 to 98.1] | 100.0 [89.4 to 100.0] | 96.9 [83.8 to 99.9] | 96.6 [82.2 to 99.9] | 92.9 [76.5 to 99.1] | 93.1 [77.2 to 99.2] | 93.5 [78.6 to 99.2] | 47.4 [24.4 to 71.1] | 61.1 [35.7 to 82.7]

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) During the Treatment Period and First 14 Follow-up Days
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE.
Time Frame: From Day 1 [post-dose] through 14 days following last dose of study drug (up to 20 weeks)
Population: All Participants as Treated (APaT) population; all randomized who received ≥1 dose of study treatment according to treatment actually received. One participant randomized to A3 arm was treated on A2 arm and thus was counted under the A2 arm (n=28).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 25 | 28 | 12 | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21
percentage of participants | 88.0 [68.8 to 97.5] | 85.7 [67.3 to 96.0] | 91.7 [61.5 to 99.8] | 90.0 [73.5 to 97.9] | 72.7 [54.5 to 86.7] | 87.1 [70.2 to 96.4] | 77.4 [58.9 to 90.4] | 65.5 [45.7 to 82.1] | 87.5 [71.0 to 96.5] | 83.9 [66.3 to 94.5] | 81.3 [63.6 to 92.8] | 78.8 [61.1 to 91.0] | 97.0 [84.2 to 99.9] | 81.3 [63.6 to 92.8] | 65.5 [45.7 to 82.1] | 53.3 [34.3 to 71.7] | 73.3 [54.1 to 87.7] | 54.8 [36.0 to 72.7] | 85.0 [62.1 to 96.8] | 90.5 [69.6 to 98.8]

3. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to an AE During the Treatment Period and First 14 Follow-up Days
Description: as for outcome 2
Time Frame: From Day 1 [post-dose] through 14 days following last dose of study drug (up to 20 weeks)
Population: APaT population; all randomized who received ≥1 dose of study treatment according to treatment actually received. One participant randomized to A3 arm was treated on A2 arm and thus was counted under the A2 arm (n=28).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 25 | 28 | 12 | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21
percentage of participants | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 10.6] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.9] | 6.3 [0.8 to 20.8] | 0.0 [0.0 to 11.2] | 3.1 [0.1 to 16.2] | 0.0 [0.0 to 10.6] | 0.0 [0.0 to 10.6] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 16.8] | 4.8 [0.1 to 23.8]

4. Secondary Outcome: Mean Time to First Achievement of Undetectable Hepatitis C Virus Ribonucleic Acid (HCV RNA)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. Kaplan Meier summary statistics were used to characterize the time to first achievement of undetectable HCV RNA.
Time Frame: From first dose of study medication until first achievement of undetectable HCV RNA (up to 18 weeks of treatment)
Population: FAS; all randomized participants who received ≥1 dose of study treatment.
Measure: Mean (Standard Error); unit: days
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 25 | 27 | 13 | 30 | 33 | 31 | 31 | 29 | 32 | 31 | 32 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 21
days | 21.7 (2.2) | 19.2 (1.8) | 23.4 (2.9) | 27.9 (3.0) | 30.7 (2.3) | 32.0 (3.0) | 37.0 (2.8) | 33.2 (2.4) | 33.1 (2.8) | 33.7 (2.6) | 31.9 (2.2) | 37.4 (2.5) | 37.4 (2.7) | 42.7 (3.3) | 27.6 (3.0) | 29.0 (2.9) | 23.7 (2.1) | 34.5 (2.6) | 30.1 (3.7) | 19.8 (2.3)

5. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA at Week 2
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. Undetectable HCV RNA was defined as below the 15.1 IU/ml limit of detection. The percentage of participants achieving undetectable HCV RNA and accompanying 95% CIs were reported at TW2 for each treatment arm of the PP Population. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 2
Population: The PP population; all randomized participants who received ≥1 dose of study treatment and without important protocol deviations who had data available at the respective time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 23 | 25 | 12 | 29 | 30 | 31 | 30 | 29 | 32 | 31 | 31 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 20
percentage of participants | 52.2 [30.6 to 73.2] | 44.0 [24.4 to 65.1] | 41.7 [15.2 to 72.3] | 44.8 [26.4 to 64.3] | 20.0 [7.7 to 38.6] | 16.1 [5.5 to 33.7] | 6.7 [0.8 to 22.1] | 10.3 [2.2 to 27.4] | 25.0 [11.5 to 43.4] | 16.1 [5.5 to 33.7] | 12.9 [3.6 to 29.8] | 6.1 [0.7 to 20.2] | 6.1 [0.7 to 20.2] | 6.3 [0.8 to 20.8] | 37.9 [20.7 to 57.7] | 40.0 [22.7 to 59.4] | 46.7 [28.3 to 65.7] | 12.9 [3.6 to 29.8] | 40.0 [19.1 to 63.9] | 70.0 [45.7 to 88.1]

6. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA at Week 4
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. Undetectable HCV RNA was defined as below the 15.1 IU/ml limit of detection. The percentage of participants achieving undetectable HCV RNA and accompanying 95% CIs were reported at TW4 for each treatment arm of the PP Population. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 4
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 23 | 24 | 12 | 30 | 30 | 31 | 30 | 29 | 32 | 31 | 30 | 32 | 33 | 32 | 29 | 28 | 30 | 31 | 20 | 18
percentage of participants | 73.9 [51.6 to 89.8] | 91.7 [73.0 to 99.0] | 75.0 [42.8 to 94.5] | 73.3 [54.1 to 87.7] | 83.3 [65.3 to 94.4] | 77.4 [58.9 to 90.4] | 60.0 [40.6 to 77.3] | 79.3 [60.3 to 92.0] | 71.9 [53.3 to 86.3] | 71.0 [52.0 to 85.8] | 83.3 [65.3 to 94.4] | 68.8 [50.0 to 83.9] | 69.7 [51.3 to 84.4] | 53.1 [34.7 to 70.9] | 75.9 [56.5 to 89.7] | 78.6 [59.0 to 91.7] | 86.7 [69.3 to 96.2] | 74.2 [55.4 to 88.1] | 50.0 [27.2 to 72.8] | 77.8 [52.4 to 93.6]

7. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA at Week 12
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. Undetectable HCV RNA was defined as below the 15.1 IU/ml limit of detection. The percentage of participants achieving undetectable HCV RNA and accompanying 95% CIs were reported at TW12 for each treatment arm of the PP Population (as applicable). 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 12
Population: The PP population; all randomized participants who received ≥1 dose of study treatment and without important protocol deviations who had data available at the respective time point. The B1, C1, and C2 arms only received 8 weeks of treatment and were thus excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 22 | 24 | 12 | 0 | 29 | 31 | 30 | 29 | 31 | 31 | 30 | 32 | 33 | 32 | 29 | 28 | 0 | 0 | 19 | 20
percentage of participants | 100.0 [84.6 to 100.0] | 100.0 [85.8 to 100.0] | 100.0 [73.5 to 100.0] |  | 100.0 [88.1 to 100.0] | 100.0 [88.8 to 100.0] | 93.3 [77.9 to 99.2] | 96.6 [82.2 to 99.9] | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [88.4 to 100.0] | 93.8 [79.2 to 99.2] | 100.0 [89.4 to 100.0] | 96.9 [83.8 to 99.9] | 93.1 [77.2 to 99.2] | 92.9 [76.5 to 99.1] |  |  | 47.7 [24.4 to 71.1] | 65.0 [40.8 to 84.6]

8. Secondary Outcome: Percentage of Participants Achieving HCV RNA <25 IU/mL at Week 2
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a LLoQ of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). The percentage of participants achieving HCV RNA levels <25 IU/ml and accompanying 95% CIs were reported at TW2 for each treatment arm of the PP Population. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 23 | 25 | 12 | 29 | 30 | 31 | 30 | 29 | 32 | 31 | 31 | 33 | 33 | 32 | 29 | 30 | 30 | 31 | 20 | 20
percentage of participants | 91.3 [72.0 to 98.9] | 92.0 [74.0 to 99.0] | 91.7 [61.5 to 99.8] | 86.2 [68.3 to 96.1] | 73.3 [54.1 to 87.7] | 77.4 [58.9 to 90.4] | 60.0 [40.6 to 77.3] | 79.3 [60.3 to 92.0] | 78.1 [60.0 to 90.7] | 67.7 [48.6 to 83.3] | 77.4 [58.9 to 90.4] | 66.7 [48.2 to 82.0] | 57.6 [39.2 to 74.5] | 62.5 [43.7 to 78.9] | 89.7 [72.6 to 97.8] | 76.7 [57.7 to 90.1] | 76.7 [57.7 to 90.1] | 61.3 [42.2 to 78.2] | 70.0 [45.7 to 88.1] | 85.0 [62.1 to 96.8]

9. Secondary Outcome: Percentage of Participants Achieving HCV RNA <25 IU/mL at Week 4
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a LLoQ of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). The percentage of participants achieving HCV RNA levels <25 IU/ml and accompanying 95% CIs were reported at TW4 for each treatment arm of the PP Population. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 4
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 23 | 24 | 12 | 30 | 30 | 31 | 30 | 29 | 32 | 31 | 30 | 32 | 33 | 32 | 29 | 28 | 30 | 31 | 20 | 18
percentage of participants | 100.0 [85.2 to 100.0] | 100.0 [85.8 to 100.0] | 100.0 [73.5 to 100.0] | 100.0 [88.4 to 100.0] | 100.0 [88.4 to 100.0] | 100.0 [88.8 to 100.0] | 90.0 [73.5 to 97.9] | 100.0 [88.1 to 100.0] | 100.0 [89.1 to 100.0] | 90.3 [74.2 to 98.0] | 100.0 [88.4 to 100.0] | 96.9 [83.8 to 99.9] | 97.0 [84.2 to 99.9] | 93.8 [79.2 to 99.2] | 100.0 [88.1 to 100.0] | 100.0 [87.7 to 100.0] | 100.0 [88.4 to 100.0] | 96.8 [83.3 to 99.9] | 65.0 [40.8 to 84.6] | 83.3 [58.6 to 96.4]

10. Secondary Outcome: Percentage of Participants Achieving HCV RNA <25 IU/mL at Week 12
Description: HCV-RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test (v.2.0) on blood samples drawn from each participant during treatment at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a LLoQ of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). The percentage of participants achieving HCV RNA levels <25 IU/ml and accompanying 95% CIs were reported at TW12 for each treatment arm of the PP Population (as applicable). 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: Week 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 22 | 24 | 12 | 0 | 29 | 31 | 30 | 29 | 31 | 31 | 30 | 32 | 33 | 32 | 29 | 28 | 0 | 0 | 19 | 20
percentage of participants | 100.0 [84.6 to 100.0] | 100.0 [85.8 to 100.0] | 100.0 [73.5 to 100.0] |  | 100.0 [88.1 to 100.0] | 100.0 [88.8 to 100.0] | 93.3 [77.9 to 99.2] | 100.0 [88.1 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [88.4 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [89.4 to 100.0] | 96.9 [83.8 to 99.9] | 100.0 [88.1 to 100.0] | 92.9 [76.5 to 99.1] |  |  | 47.4 [24.4 to 71.1] | 75.0 [50.9 to 91.3]

11. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 4 Weeks After the End of All Therapy (SVR4)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a LLoQ of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). SVR4 was defined as HCV RNA <25 IU/ml at 4 weeks after the end of all study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: 4 weeks after end of therapy (up to 22 weeks)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 22 | 24 | 12 | 30 | 29 | 31 | 30 | 29 | 31 | 31 | 30 | 33 | 33 | 32 | 29 | 29 | 29 | 31 | 20 | 18
percentage of participants | 100.0 [84.6 to 100.0] | 95.8 [78.9 to 99.9] | 100.0 [73.5 to 100.0] | 93.3 [77.9 to 99.2] | 100.0 [88.1 to 100.0] | 96.8 [83.3 to 99.9] | 96.7 [82.8 to 99.9] | 96.6 [82.2 to 99.9] | 100.0 [88.8 to 100.0] | 96.8 [83.3 to 99.9] | 100.0 [88.4 to 100.0] | 93.9 [79.8 to 99.3] | 100.0 [89.4 to 100.0] | 96.9 [83.8 to 99.9] | 96.6 [82.2 to 99.9] | 93.1 [77.2 to 99.2] | 93.1 [77.2 to 99.2] | 96.8 [83.3 to 99.9] | 50.0 [27.2 to 72.8] | 61.1 [35.7 to 82.7]

12. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of All Study Therapy (SVR24)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 at various time points prior to, during, and after dosing. The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a LLoQ of 25 IU/mL and a limit of detection of 15.1 IU/mL (in plasma). SVR24 was defined as HCV RNA <25 IU/ml at 24 weeks after the end of all study therapy. 95% confidence intervals provided based on the Clopper-Pearson method.
Time Frame: 24 weeks after end of therapy (up to 42 weeks)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Number analyzed (Participants) | 20 | 24 | 12 | 28 | 29 | 31 | 30 | 29 | 31 | 29 | 29 | 33 | 32 | 32 | 29 | 27 | 29 | 31 | 19 | 17
percentage of participants | 100.0 [83.2 to 100.0] | 95.8 [78.9 to 99.9] | 100.0 [73.5 to 100.0] | 78.6 [59.0 to 91.7] | 100.0 [88.1 to 100.0] | 96.8 [83.3 to 99.9] | 90.0 [73.5 to 97.9] | 96.6 [82.2 to 99.9] | 100.0 [88.8 to 100.0] | 93.1 [77.2 to 99.2] | 100.0 [88.1 to 100.0] | 90.9 [75.7 to 98.1] | 100.0 [89.1 to 100.0] | 96.9 [83.8 to 99.9] | 96.6 [82.2 to 99.9] | 88.9 [70.8 to 97.6] | 93.1 [77.2 to 99.2] | 93.5 [78.6 to 99.2] | 47.4 [24.4 to 71.1] | 58.8 [32.9 to 81.6]

ADVERSE EVENTS:
Time Frame: Treatment and Follow-up periods (up to 42 weeks)
Description: All Participants as Treated (APaT) population; all randomized who received ≥1 dose of study treatment according to treatment actually received. One participant randomized to A3 arm was treated on A2 arm and thus was counted under the A2 arm (n=28).
Arm/Group | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/28 | 0/12 | 0/30 | 0/33 | 0/31 | 1/31 | 2/29 | 1/32 | 1/31 | 2/32 | 1/33 | 0/33 | 1/32 | 1/29 | 2/30 | 1/30 | 0/31 | 0/20 | 2/21
Other Adverse Events (participants affected / at risk) | 19/25 | 24/28 | 11/12 | 27/30 | 23/33 | 24/31 | 23/31 | 18/29 | 26/32 | 24/31 | 24/32 | 25/33 | 32/33 | 25/32 | 18/29 | 14/30 | 22/30 | 14/31 | 16/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk (N=25) | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=28) | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=12) | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=30) | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=33) | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=31) | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=31) | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk (N=29) | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (N=32) | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk (N=31) | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk (N=32) | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=33) | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=33) | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk (N=32) | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=29) | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=30) | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=30) | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk (N=31) | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=20) | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (N=21)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: TN NC Grazoprevir 100 mg + Elbasvir 20 mg + RBV-12 wk (N=25) | A2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=28) | A3: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=12) | B1: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=30) | B2: TN NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=33) | B3: TN NC/GT1a Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=31) | B4: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=31) | B5: TN C Grazoprevir 100 mg + Elbasvir 50 mg for 12 wk (N=29) | B6: TN C Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (N=32) | B7: TN C Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk (N=31) | B8: NR Grazoprevir 100 mg + Elbasvir 50 mg +RBV-12 wk (N=32) | B9: NR Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=33) | B10: NR Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=33) | B11: NR Grazoprevir 100 mg + Elbasvir 50 Mg-18 wk (N=32) | B12: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=29) | B13: TN HIV NC Grazoprevir 100 mg + Elbasvir 50 Mg-12 wk (N=30) | C1: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 mg + RBV-8 wk (N=30) | C2: TN NC/GT1b Grazoprevir 100 mg + Elbasvir 50 Mg-8 wk (N=31) | D1: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-12 wk (N=20) | D2: TN NC/GT3 Grazoprevir 100 mg + Elbasvir 50 mg + RBV-18 wk (N=21)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1) | 5 (5) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7) | 2 (2) | 8 (8) | 6 (6) | 5 (5) | 4 (4) | 0 (0) | 4 (5) | 4 (5) | 4 (4) | 2 (2) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 3 (3) | 3 (3) | 6 (7)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (5) | 2 (2) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 5 (6) | 2 (2) | 7 (7) | 5 (7) | 6 (6) | 7 (7) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 5 (5) | 4 (4) | 15 (15) | 10 (10) | 6 (7) | 11 (11) | 6 (6) | 9 (10) | 6 (7) | 6 (6) | 10 (12) | 15 (16) | 8 (8) | 2 (2) | 2 (2) | 11 (11) | 3 (3) | 2 (2) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 5 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 2 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 3 (4) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 6 (6) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 5 (5) | 7 (7) | 7 (9) | 10 (11) | 2 (3) | 4 (5) | 11 (13) | 10 (12) | 10 (12) | 6 (6) | 6 (7) | 10 (10) | 4 (5) | 2 (2) | 6 (6) | 5 (6) | 5 (5) | 5 (5)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 7 (8) | 2 (2) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 2 (3) | 3 (3) | 6 (6) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Irritability (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 5 (5) | 1 (1) | 5 (6) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 6 (6) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 10 (10) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 7 (8) | 0 (0) | 3 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (6) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.